CLINICAL TRIAL: NCT00216398
Title: A Phase IV, Open-label, Single Group Study to Evaluate the Dosing, Efficacy and Safety of Lanreotide Autogel® in Patients With Acromegaly Previously Treated With Octreotide LAR
Brief Title: Lanreotide Autogel in Patients With Acromegaly Previously Treated With Octreotide LAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-9B-52030-159
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
Keywords: acromegaly; growth hormone
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation)

SUMMARY:
The purpose of this study is to assess the efficacy, safety and patient acceptability of Somatuline Autogel in patients with acromegaly previously treated with octreotide LAR.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acromegaly
* The patient must have been tested at Week -4 (4 weeks prior to the Baseline visit) and shown to have a GH level <10 mU/L.
* The patient must have been treated with a stable dose of octreotide LAR for at least four months prior to study entry
* Life expectancy of at least 2 years

Exclusion Criteria:

* Adenectomy within past 6 months, or likely during study period
* Radiotherapy for acromegalic disease within 1 year, or likely during study period
* Unstable concomitant dopamine agonist therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06-22 (Actual); Study Completion 2006-06-22 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with GH control (<5.0 mU.L) and normalised IGF-1 at week 44 compared to the baseline (Week 0) visit.

SECONDARY OUTCOMES:
The percentage of patients with GH control (< 5.0 mU/L) at each visit to week 44 compared to the baseline (Week 0) visit.
The percentage of patients with normalised IGF-1 compared to the baseline visit.
Change in the GH values compared to the baseline (Week 0) visit.
Change in the IGF-1 values compared to the baseline (Week 0) visit.
Change in serum lanreotide levels compared to the baseline (Week 0) visit.
Change in the serum octreotide levels compared to the baseline visit.
Patient evaluation of lanreotide Autogel treatment compared with evaluation of octreotide LAR treatment.
Investigator evaluation of lanreotide Autogel treatment compared with evaluation of octreotide LAR treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia